CLINICAL TRIAL: NCT00485979
Title: A Randomized, Open-label, Multi-center Study of Larotaxel at 90mg/m2 or Docetaxel Every 3 Weeks, Alone or in Combination With Trastuzumab According to Her2neu Status, Administered After a Combination of Anthracycline and Cyclophosphamide as Pre-operative Therapy in Patients With High Risk Localized Breast Cancer.
Brief Title: Treatment of Larotaxel/Docetaxel, +/- Trastuzumab, After Anthracycline-cyclophosphamide in Breast Cancer Patients
Acronym: SATIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC10073; EudraCT 2006-006473-24
Record Dates: First submitted 2007-06-12; First posted 2007-06-13 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer; Neoadjuvant therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — larotaxel; Docetaxel; Trastuzumab

ARMS (4):
- Arm A1 (Experimental): Cohort 1: Her2-ve breast cancer
  Interventions: Drug: larotaxel (XRP9881)
- Arm B1 (Active Comparator): Cohort 1: Her2-ve breast cancer
  Interventions: Drug: docetaxel
- Arm A2 (Experimental): Cohort 2: Her2+ve breast cancer
  Interventions: Drug: larotaxel (XRP9881); Drug: trastuzumab
- Arm B2 (Active Comparator): Cohort 2: Her2+ve breast cancer
  Interventions: Drug: docetaxel; Drug: trastuzumab

INTERVENTIONS:
Drug: larotaxel (XRP9881) — intravenous administration
  Arms: Arm A1; Arm A2
Drug: docetaxel — intravenous administration
  Arms: Arm B1; Arm B2
Drug: trastuzumab — intravenous administration
  Arms: Arm A2; Arm B2

SUMMARY:
The primary objective of this study is to assess the pathological Complete Response (pCR) rate by treatment arm (according to Chevallier criteria).

The secondary objectives are:

* to assess in each treatment arm the clinical Response Rate (RR), the rate of breast conservation, the Progression-Free Survival (PFS), the Overall Survival (OS), the safety and tolerability profile, the pathological Complete Response rate (pCR) according to NSABP and Sataloff criteria,
* to rank docetaxel and larotaxel alone in Her2 -ve patients, or combined with trastuzumab in Her2 +ve patients, according to the pCR rate.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven invasive breast adenocarcinoma
* Localized breast cancer: stage II and III
* Tumors clinically palpable and ineligible for breast conservative surgery: unifocal tumor with diameter ≥ 3cm (clinical examination) or central unifocal tumor, or whose characteristics make pre-operative chemotherapy mandatory due to high risk factors (i.e. ipsilateral lymph nodes involvement, rapid growth rate)
* After 30 June 2008, known status for Her2neu by immunohistochemistry (IHC) or by fluorescent in situ hybridization (FISH)

Exclusion Criteria:

* Bilateral and inflammatory breast cancer
* Abnormal Left Ventricular Ejection Fraction
* Distant metastases or locoregional relapse
* Inadequate organ functions

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2007-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Pathological response will be assessed according to Chevallier criteria for patients who underwent surgery. | treatment period

SECONDARY OUTCOMES:
Clinical Response Rate, Rate of breast conservation, Progression-Free Survival, Overall Survival, pathological response according to NSABP and Sataloff criteria for patients who underwent surgery | treatment period
Safety and tolerability profile | treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Michel Marty, MD, Principal Investigator — Centre for Therapeutic Innovations in Oncology and Haematology / Saint Louis University Hospital
Locations (8):
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Mégrine, Tunisia
- Sanofi-Aventis Administrative Office, Guildford, United Kingdom
- Sanofi-Aventis Administrative Office, Montevideo, Uruguay